CLINICAL TRIAL: NCT03915782
Title: NeuroPRotective Effect of remOte Ischemic condiTioning in Ischemic strokE Treated With meChanical Thrombectomy (PROTECT-I Study)
Brief Title: Neuroprotective Effect of Remote Ischemic Conditioning in Ischemic Stroke Treated With Mechanical Thrombectomy
Acronym: PROTECT-I
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 69HCL19_0129; 2019-A01052-55 (Other: ID-RCB)
Record Dates: First submitted 2019-04-11; First posted 2019-04-16 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Stroke, Ischemic
Keywords: Ischemic stroke; Mechanical Thrombectomy; Ischemia/Reperfusion; Remote Ischemic Conditioning; Magnetic Resonance Imaging
MeSH Terms: conditions — Ischemic Stroke; Ischemia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remote Ischemic Conditioning (RIC) positive (Experimental): Patients with remote ischemic conditioning
  Interventions: Device: Remote ischemic conditioning
- Control group (Sham Comparator): The control group will receive a sham procedure (same procedure than Remote Ischemic Conditioning (RIC) with brachial cuff inflation to 30 millimeters (mm) of mercury (Hg) during 40 minutes).
  Interventions: Device: Patients with a sham procedure of remote ischemic conditioning

INTERVENTIONS:
Device: Remote ischemic conditioning — Remote ischemic conditioning (RIC): Four cycles of [5 minutes of brachial cuff inflation at 200 millimeters (mm) of mercury (Hg) followed by 5 minutes of cuff deflation] started as soon as possible after Magnetic Resonance Imaging (MRI).
  Arms: Remote Ischemic Conditioning (RIC) positive
Device: Patients with a sham procedure of remote ischemic conditioning — Sham procedure: Four cycles of [5 minutes of brachial cuff inflation at 30 millimeters (mm) of mercury (Hg) followed by 5 minutes of cuff deflation] started as soon as possible after Magnetic Resonance Imaging (MRI).
  Arms: Control group

SUMMARY:
The benefit of mechanical thrombectomy in the treatment of ischemic stroke has been demonstrated in several multicenter randomized trials. However, it leads to a sudden reperfusion of the brain parenchyma associated to an extension of the infarct volume. Evidence has indicated that remote ischemic conditioning (RIC) reduces final infarct size in animal stroke models. The main objective of the present study is to determine whether remote ischemic conditioning can limit the final infarct volume after recanalization of the occluded cerebral artery.

ELIGIBILITY:
Inclusion Criteria:

* Age at least 18 years old,
* Carotid ischemic stroke related to a full occlusion of the middle cerebral artery (occlusion of middle 1 (M1) and/or proximal middle 2 (M2) identified as candidate for endovascular intervention according to local criteria,
* Brain Magnetic Resonance Imaging (MRI) performed within 6 hours from symptoms onset,
* Acute stroke MRI including at least diffusion weighted imaging (DWI), fluid attenuated inversion recovery (FLAIR), intracranial vessel imaging with Magnetic Resonance Angiography (MRA) and perfusion weighted imaging (PWI),
* Modified Rankin Score (mRS) score less than or equal to 1 before ischemic stroke,
* Obtaining a written informed consent of the patient or a next of kin, or emergency inclusion process.

Non inclusion Criteria:

* Previous ischemic stroke or transient ischemic attack (TIA) in the previous 3 months,
* Contraindications to iodinated contrast agents,
* Sickle cell disease known (risk of vaso-occlusive crisis),
* Life expectancy less than 90 days,
* Pregnant or women of childbearing age who were not using contraception (oral diagnosis),
* Patient without health coverage,
* Patient under legal protection.
* Any contraindication to Magnetic Resonance Imaging (MRI) (example cardiac pacemaker),
* Intracranial bleeding,
* Intracranial expansive process.

Exclusion Criteria:

* Recanalization of M1 or proximal M2 segment at the time of thrombectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2020-03-20 (Actual); Primary Completion 2024-07-11 (Actual); Study Completion 2024-10-21 (Actual)

PRIMARY OUTCOMES:
Final volume of cerebral infarction measured by Magnetic Resonance Imaging (MRI) at Day 1 after thrombectomy | Day 1 after thrombectomy
  Measurement of the final volume of cerebral infarction on Fluid Attenuated Inversion Recovery (FLAIR) sequence by a blinding imaging reading committee.

SECONDARY OUTCOMES:
Change in Neurological prognosis | 1/ National Institutes of Health Stroke Scale (NIHSS) score will be evaluated at day 7; 2/ Modified Rankin Score (mRS) will be evaluated at day 90 and 3/ Incidence of early neurological worsening will be evaluated at inclusion and up to day 1.
  Functional neurological prognosis assessed by: 1/ National Institutes of Health Stroke Scale (NIHSS) score on day 7 (NIHSS score for each ability is a number between 0 and 4 with 0 being normal functioning and 4 being completely impaired. The patient's NIHSS score is calculated by adding the number for each element of the scale; 42 is the highest score possible. The higher the score, the more impaired neurologically a stroke patient is) 2/ Modified Rankin Score (MRS) score at 90 days (score from 0 to 6 with 0 being normal functioning and 6 being death, the higher the score the more impaired neurologically a stroke patient is) and 3/ Incidence of early neurological worsening (Difference in NIHSS score between inclusion and day 1 > 4 points).
Change in growth of the supposed irreversible lesion measured by Magnetic Resonance Imaging (MRI) from admission to day 1. | Magnetic Resonance Imaging (MRI) will be performed at inclusion (Day 0) and on day 1.
  It will be expressed as a percentage of the size of the hypoperfused area measured on the admission Magnetic Resonance Imaging (MRI).
Arterial reperfusion measured by the Thrombolysis in Cerebral Infarction (TICI) score at the end of the thrombectomy procedure. | Day 1 of thrombectomy
  The Thrombolysis in Cerebral Infarction (TICI) score is a tool for determining the response of thrombolytic therapy for ischemic stroke and is defined as follows: 0=no perfusion; 1= penetration, but no distal branch filling; 2a= perfusion with incomplete (<50%) distal branch filling; 2b=perfusion with incomplete (>50%) distal branch filling; and 3=full perfusion with filling of all distal branches. A score of 0 being the least favorable outcome for the patient (no perfusion) and a maximum score of 3 being the most favorable outcome for the patient (full perfusion).
Arterial reperfusion measured at Day 1 by Magnetic Resonance Imaging (MRI). | Day 1
  Arterial reperfusion according to the Arterial Occlusive Lesion (AOL) score. This score is related to recanalization of the primary arterial occlusive lesion on a scale of 0 to 3 : 0 is no recanalization of the primary occlusive lesion; 1 is incomplete or partial recanalization of the primary occlusive lesion with no distal flow; 2 is incomplete or partial recanalization of the primary lesion with any distal flow; and 3 is complete recanalization of the primary occlusive lesion with any distal flow. The most favorable outcome for the patient is a score of 3 while a score of 0 is the least favorable patient outcome.
Impact on collateral circulation assessed by the Higashida score. | Day 1
  Higashida score offers a non-invasive collateral vessel and tissue perfusion assessment of ischemic tissue. This grading system subdivides the collateral flow into five grades, from grade 0 (no collaterals visible on the ischemic side) to grade 5 (complete and rapid collateral blood flow to the vascular bed in the entire ischemic territory by retrograde perfusion). A grade of 3-5 is considered good collateral formation whereas a grade of 0-2 is considered poor collateral formation after a stroke and is less favorable to the patient's outcome.
Incidence of hemorrhagic transformation at day 1 measured by routine Magnetic Resonance Imaging (MRI) | Day 1
  European Cooperative Acute Stroke Study (ECASS) classification of potential haemorrhagic transformation which divides hemorrhagic transformation into four subtypes: 1) hemorrhagic infarction type 1 (HI1) such as petechial hemorrhages at the infarct margins; 2) hemorrhagic infarction type 2 (HI2) such as petechial hemorrhages throughout the infarct and no mass-effect attributable to the hemorrhages; 3) parenchymal hematoma type 1 (PH1) such as less than or equal to 30% of the infarcted area minor mass effect attributable to the hematoma and 4) parenchymal hematoma type 2 (PH2) such as greater than 30% of infarct zone substantial mass effect attributable to the hematoma. The most favorable patient outcome being the first classification hemorrhagic infarction type 1 (HI1) and the least favorable patient outcome being the fourth classification parenchymal hematoma type 2 (PH2).
Complications related to the endovascular procedure | Day 1
  Complications such as: embolism in an another initially not involved vascular territory, dissection, severe vasospasm that needs an intra-arterial treatment, vascular perforation
Responder analysis to thrombectomy relating Modified Rankin score (mRS) 90 days after stroke to baseline National Institutes of Health Stroke Scale (NIHSS) score. | Day 90
  NIHSS score for each ability is a number between 0 and 4 with 0 being normal functioning and 4 being completely impaired. The patient's NIHSS score is calculated by adding the number for each element of the scale; 42 is the highest score possible. The higher the score, the more impaired a stroke patient is. MRS score from 0 to 6 with 0 being normal functioning and 6 being death, the higher the score the more impaired a stroke patient is. For this study a positive response is defined by : a NIHSS <7 at admission and a MRS = 0 at Day 90 ; a NIHSS between 8 and 14 at admission and a MRS = 0 or 1 at Day 90 ; a NIHSS >14 at admission and a MRS = 0 to 2 at Day 90.

CONTACTS AND LOCATIONS:
Overall Officials: Laura MECHTOUFF, MD, Principal Investigator — Hospices Civils de Lyon, Hopital Pierre Wertheimer
Locations (1):
- Service De Neurologie Vasculaire - Hôpital Neurologique Pierre Wertheimer (GHE), Bron, France